CLINICAL TRIAL: NCT05098015
Title: Controlled Trial of Game Changers: A Group Intervention to Train HIV Clients to be Change Agents for HIV Prevention in Uganda
Brief Title: Randomized Controlled Trial of Game Changers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Infectious Diseases Institute, Uganda (Other); Makerere University (Other); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-N0155
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: HIV Prevention

STUDY DESIGN:
Intervention Model Description: Individual randomization of index participants (and their recruited alter participants) to one of two parallel groups, the intervention or usual care (no intervention) control group. Therefore there are 4 study groups: index intervention, alter intervention, index control and alter control
Who Masked: Outcomes Assessor
Masking Description: The assessment interviewer will be blinded to study arm allocation of the participants at baseline only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention- index (Experimental): 8-session group intervention to train index participants to engage in HIV prevention advocacy.
  Interventions: Behavioral: Game Changers
- Usual care control- index (No Intervention): Participants will receive HIV usual care, and no added intervention.
- Intervention- alter (No Intervention): Enrolled alter participants recruited by index participants assigned to the intervention comprise this arm
- Usual care control- alter (No Intervention): ALter participants recruited by index participants assigned to the usual care control group comprise this arm

INTERVENTIONS:
Behavioral: Game Changers — 8-session group intervention that uses didactic instruction, role plays and experience sharing to empower participants to engage in HIV prevention advocacy.
  Arms: Intervention- index

SUMMARY:
The study is a randomized controlled trial (RCT) of Game Changers, an 8-session peer-led group intervention that aims to empower and mobilize people living with HIV (PLWH) to be agents for HIV prevention in their social networks.

DETAILED DESCRIPTION:
This RCT of Game Changers, a peer-led group intervention for persons living with HIV (PLWH) in Uganda, will test intervention effects on the primary outcomes of reduced condomless sex, increased HIV testing, and decreased enacted HIV stigma among social network members. We will recruit 210 PLWH, randomizing 105 to the intervention and 105 to an attention control. Each PLWH will be asked to recruit up to 4 social network members to complete assessments (736 total, 368/arm). All participants will complete surveys at baseline and 6-, 12-, and 18-months post-baseline.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and older
* HIV-positive
* in HIV care at The Infectious DIseases Institute for at least one year

Exclusion Criteria:

* Participated in the prior pilot study of the intervention.
* Has significant cognitive impairment
* Health status is not sufficiently stable to reliably complete 18 month study.
* Does not speak Luganda fluently (index participant); English or Luganda fluently (social network participant)
* spouse/partner or household member are enrolled as index participant in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 809 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Wagner, Principal Investigator — RAND
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be made available upon review of requests from outside researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication of primary results of the study (approximately August 2026).

REFERENCES:
- [Derived] Bogart LM, Matovu JKB, Green HD Jr, Ninsiima S, Klein DJ, Gwokyalya V, Serunkuuma R, Ghosh-Dastidar B, Mubiru K, Nabukeera M, Malika N, Okoboi S, Wagner GJ. Randomized Controlled Trial of Game Changers, a Social Network Intervention for HIV Prevention in Uganda. AIDS Behav. 2025 Nov 11:10.1007/s10461-025-04907-4. doi: 10.1007/s10461-025-04907-4. Online ahead of print. PMID 41214256
- [Derived] Wagner GJ, Bogart LM, Green HD, Storholm ED, Klein DJ, McBain RK, Serunkuuma R, Mubiru K, Matovu JKB, Okoboi S. Social network-based group intervention to promote HIV prevention in Uganda: study protocol for a cluster randomized controlled trial of Game Changers. Trials. 2022 Mar 28;23(1):233. doi: 10.1186/s13063-022-06186-z. PMID 35346329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PLWH are the index participants, and each enrolled index participant was asked to recruit up to 4 social network members (alters) to also enroll in the study.
Pre-assignment Details: Both index participants (PLWH) and alter participants were enrolled; as all index participants were asked to recruit up to 4 alters, each index participant may have any where from 0 to 4 alters enrolled in the study. 210 index (PLWH) participants enrolled and 599 alters enrolled.
  The flowchart includes statistics on the number of index and alter participants enrolled and completed within each arm.
Groups:
- Intervention- Alter: Alter participants recruited by enrolled index participants assigned to receive the intervention comprise this group; however, these alter participants did not receive any intervention
- Usual Care Control- Alter: Alter participants recruited by enrolled index participants assigned to the usual care control group comprise this arm
Period: Overall Study
Arm/Group | Intervention- Index | Usual Care Control- Index | Intervention- Alter | Usual Care Control- Alter
Started | 105 | 105 | 324 | 275
Completed | 103 | 102 | 318 | 270
Not Completed | 2 | 3 | 6 | 5
Not completed — Death | 1 | 1 | 3 | 0
Not completed — Lost to Follow-up | 1 | 1 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled index and alter participants were part of analysis population
Groups:
- Usual Care Control- Alter: Alter participants recruited by enrolled index participants assigned to the usual care control group
- Intervention- Alter: Alter participants recruited by enrolled index participants assigned to the intervention group; however, these alter participants did not receive any intervention
- Total: Total of all reporting groups
Arm/Group | Intervention- Index | Usual Care Control- Index | Usual Care Control- Alter | Intervention- Alter | Total
Number analyzed (Participants) | 105 | 105 | 275 | 324 | 809
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (10.7) | 39.3 (10.5) | 38.2 (12.4) | 36.6 (12.3) | 38.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 73 | 174 | 223 | 544
  Male | 31 | 32 | 101 | 101 | 265
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 105 | 105 | 275 | 324 | 809
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Time since HIV diagnosis [Mean (Standard Deviation); unit: years] — Population: This measure was only assessed among index participants (in both the intervention-index and usual care control-index arms), all of whom were persons living with HIV
  years
    number analyzed (Participants) | 105 | 105 | 0 | 0 | 210
    (all) | 10.8 (6.1) | 11.1 (5.2) |  |  | 11.0 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: HIV Testing
Description: For each index participant (PLWH), data is examined from their enrolled alters and the percent of these alters who self-reported HIV testing behavior (yes/no) at each follow-up assessment is calculated, followed by the average percent across all follow-up assessments. Therefore, data from all three follow-up timepoints (months 6, 12 18) were pooled and an average calculated across the timepoints.
Time Frame: Data regarding HIV testing over the past 6 months, assessed at each follow-up assessment (Months 6, 12, 18)
Population: The Participant Flow included data from all index (PLWH) and alter participants, while the outcome measures are based on index-level measures-- for each index participant, the measure reflects data reported by their enrolled alters. For this specific measure (HIV testing), index participants provided data for analysis if (a) at least one of their alters was not living with HIV at the time of the assessment; and (2) data was present in at least one of the follow-up assessments
Measure: Mean (Standard Deviation); unit: percentage of alters
Groups:
- Intervention- Index: 8-session group intervention to train participants to engage in HIV prevention advocacy.
  Game Changers: 8-session group intervention that uses didactic instruction, role plays and experience sharing to empower participants to engage in HIV prevention advocacy.
Arm/Group | Intervention- Index | Usual Care Control- Index
Number analyzed (Participants) | 91 | 78
percentage of alters | 71.60 (35.23) | 71.61 (37.19)
Statistical Analysis 1: Comparison: Intervention- Index vs Usual Care Control- Index; Test type: Superiority; p = 0.95, Regression, Linear; Slope = 0.25, Standard Error of Mean 4.16

2. Primary Outcome: Condom Use
Description: For each index participant (PLWH), data is examined from their enrolled alters and the percent of these alters who self-reported always using condoms use during intercourse at each follow-up assessment is calculated, followed by the average percentage across all follow-up assessments. Therefore, data from all three follow-up timepoints (months 6, 12 18) were pooled and an average calculated across the timepoints.
Time Frame: Reports of always using condoms in the past 6 months, as assessed at each follow-up assessment (Month 6, Month 12, Month 18)
Population: The Participant Flow included data from all index (PLWH) and alter participants, while the outcome measures are based on index-level measures-- for each index participant, the measure reflects data reported by their enrolled alters. Index participants were included in the analysis if (a) at least one of their alters reported engaging in sexual intercourse in the 6 months prior to the assessment; and (b) data was available in at least one of the follow-up assessments
Measure: Mean (Standard Deviation); unit: percentage of alters
Groups:
- Intervention: 8-session group intervention to train participants to engage in HIV prevention advocacy.
  Game Changers: 8-session group intervention that uses didactic instruction, role plays and experience sharing to empower participants to engage in HIV prevention advocacy.
- Usual Care Control: Participants will receive HIV usual care, and no added intervention.
Arm/Group | Intervention | Usual Care Control
Number analyzed (Participants) | 92 | 88
percentage of alters | 18.04 (29.60) | 13.15 (27.06)
Statistical Analysis 1: Comparison: Intervention vs Usual Care Control; Test type: Superiority; p = 0.16, Regression, Linear; Slope = 4.38, Standard Error of Mean 3.12

3. Secondary Outcome: Internalized HIV Stigma
Description: This outcome is based solely on data from the index participants. Self-reported internalized HIV stigma (on 1-5 scale, with higher scores represented greater stigma); scale score is averaged across all follow-up assessments
Time Frame: Reported at each follow-up assessment (Months 6, 12, 18)
Population: The Participant Flow included data from all index (PLWH) and alter participants, but this measure was only assessed among index participants. Index participants were included in the analysis if they provided data on the measure in at least one follow-up assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention- Index | Usual Care Control- Index
Number analyzed (Participants) | 105 | 104
score on a scale | 1.62 (0.72) | 2.06 (0.91)
Statistical Analysis 1: Comparison: Intervention- Index vs Usual Care Control- Index; Test type: Superiority; p < .001, Regression, Linear; Slope = -0.46, Standard Error of Mean 0.08

4. Secondary Outcome: HIV Prevention Advocacy
Description: This outcome is based solely on data from the index participants. Self-reported prevention advocacy (on 1-5 scale, with higher scores representing greater engagement in advocacy); scores are averaged across all follow-up assessments
Time Frame: Past 6 months as assessed at each follow-up (Months 6, 12, 18)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention- Index | Usual Care Control- Index
Number analyzed (Participants) | 105 | 104
score on a scale | 3.53 (0.91) | 2.85 (1.05)
Statistical Analysis 1: Comparison: Intervention- Index vs Usual Care Control- Index; Test type: Superiority; p < .001, Regression, Linear; Slope = 0.67, Standard Error of Mean 0.10

ADVERSE EVENTS:
Time Frame: Each participant was assessed over 18 months from enrollment.
Description: Adverse events were assessed for all index (PLWH) and alter participants.
Groups:
- Intervention- Alter: Alter participants recruited by index participants assigned to the intervention group comprise this arm; however, these alter participants did not receive an intervention
Arm/Group | Intervention- Index | Usual Care Control- Index | Usual Care Control- Alter | Intervention- Alter
All-Cause Mortality (participants affected / at risk) | 1/105 | 1/105 | 0/275 | 3/324
Serious Adverse Events (participants affected / at risk) | 2/105 | 0/105 | 0/275 | 0/324
Other Adverse Events (participants affected / at risk) | 0/105 | 0/105 | 0/275 | 0/324
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention- Index (N=105) | Usual Care Control- Index (N=105) | Usual Care Control- Alter (N=275) | Intervention- Alter (N=324)
domestic violence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
loss of job (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT05098015/Prot_SAP_000.pdf